CLINICAL TRIAL: NCT05765838
Title: Combined Molecular Testing for Influenza, SARS-CoV-2, and RSV RNA From Different Upper Airway Specimens.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tobias Todsen, MD, Phd, Consultant, Ass. Prof, Rigshospitalet, Denmark
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: H-23006949
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Influenza; COVID-19; RSV Infection
MeSH Terms: conditions — Influenza, Human; COVID-19; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: The order of the swabs performed will be decided with randomization to either of the eight combination:
  1. NPS right - Nasal swab left - OPS
  2. NPS left - Nasal swab right - OPS
  3. Nasal swab right - NPS left - OPS
  4. Nasal swab left - NPS right - OPS
  5. NPS right - OPS - Nasal swab left
  6. NPS left - OPS - Nasal swab right
  7. Nasal swab right - OPS - NPS left
  8. Nasal swab left - OPS - NPS right
  9. OPS - NPS right - Nasal swab left
  10. OPS - NPS left - Nasal swab right
  11. OPS - Nasal swab left - NPS right
  12. OPS - Nasal swab right - NPS left
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Sequence for upper airway specimen collection (NPS right - Nasal swab left - OPS) (Experimental): 1 NPS right - Nasal swab left - OPS
  NPS = nasopharyngeal swab OPS = oropharyngeal swab
  Interventions: Diagnostic Test: (NPS right - Nasal swab left - OPS)
- Sequence for upper airway specimen collection (NPS left - Nasal swab right - OPS) (Experimental): 2 NPS left - Nasal swab right - OPS
  Interventions: Diagnostic Test: (NPS left - Nasal swab right - OPS)
- Sequence for upper airway specimen collection (Nasal swab right - NPS left - OPS) (Experimental): 3 Nasal swab right - NPS left - OPS
  Interventions: Diagnostic Test: (Nasal swab right - NPS left - OPS)
- Sequence for upper airway specimen collection (Nasal swab left - NPS right - OPS) (Experimental): 4 Nasal swab left - NPS right - OPS
  Interventions: Diagnostic Test: (Nasal swab left - NPS right - OPS)
- Sequence for upper airway specimen collection (NPS right - OPS - Nasal swab left) (Experimental): 5 NPS right - OPS - Nasal swab left
  Interventions: Diagnostic Test: (NPS right - OPS - Nasal swab left)
- Sequence for upper airway specimen collection (NPS left - OPS - Nasal swab right) (Experimental): 6 NPS left - OPS - Nasal swab right
  Interventions: Diagnostic Test: (NPS left - OPS - Nasal swab right)
- Sequence for upper airway specimen collection (Nasal swab right - OPS - NPS left) (Experimental): 7 Nasal swab right - OPS - NPS left
  Interventions: Diagnostic Test: (Nasal swab right - OPS - NPS left)
- Sequence for upper airway specimen collection (Nasal swab left - OPS - NPS right) (Experimental): 8 Nasal swab left - OPS - NPS right
  Interventions: Diagnostic Test: (Nasal swab left - OPS - NPS right)
- Sequence for upper airway specimen collection (OPS - NPS right - Nasal swab left) (Experimental): 9 OPS - NPS right - Nasal swab left
  Interventions: Diagnostic Test: (OPS - NPS right - Nasal swab left)
- Sequence for upper airway specimen collection (OPS - NPS left - Nasal swab right) (Experimental): 10 OPS - NPS left - Nasal swab right
  Interventions: Diagnostic Test: (OPS - NPS left - Nasal swab right)
- Sequence for upper airway specimen collection (OPS - Nasal swab left - NPS right) (Experimental): 11 OPS - Nasal swab left - NPS right
  Interventions: Diagnostic Test: (OPS - Nasal swab left - NPS right)
- Sequence for upper airway specimen collection (OPS - Nasal swab right - NPS left) (Experimental): 12 OPS - Nasal swab right - NPS left
  Interventions: Diagnostic Test: (OPS - Nasal swab right - NPS left)

INTERVENTIONS:
Diagnostic Test: (NPS right - Nasal swab left - OPS) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (NPS right - Nasal swab left - OPS)
Diagnostic Test: (NPS left - Nasal swab right - OPS) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (NPS left - Nasal swab right - OPS)
Diagnostic Test: (Nasal swab right - NPS left - OPS) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (Nasal swab right - NPS left - OPS)
Diagnostic Test: (Nasal swab left - NPS right - OPS) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (Nasal swab left - NPS right - OPS)
Diagnostic Test: (NPS right - OPS - Nasal swab left) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (NPS right - OPS - Nasal swab left)
Diagnostic Test: (NPS left - OPS - Nasal swab right) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (NPS left - OPS - Nasal swab right)
Diagnostic Test: (Nasal swab right - OPS - NPS left) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (Nasal swab right - OPS - NPS left)
Diagnostic Test: (Nasal swab left - OPS - NPS right) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (Nasal swab left - OPS - NPS right)
Diagnostic Test: (OPS - NPS right - Nasal swab left) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (OPS - NPS right - Nasal swab left)
Diagnostic Test: (OPS - NPS left - Nasal swab right) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (OPS - NPS left - Nasal swab right)
Diagnostic Test: (OPS - Nasal swab left - NPS right) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (OPS - Nasal swab left - NPS right)
Diagnostic Test: (OPS - Nasal swab right - NPS left) — Collection of nasopharyngeal-, nasal-, and oropharyngeal swabs in randomized order
  Arms: Sequence for upper airway specimen collection (OPS - Nasal swab right - NPS left)

SUMMARY:
This is a comparative prospective diagnostic accuracy study reported according to the STARD guidelines. Citizens at an outpatient COVID19 test facility at Testcenter Danmark Valby will be invited to participate in the study on a volunteer basis. The enrolled participants will have the planned oropharyngeal swab performed in the test center and sent for a SARS-CoV-2 RT-PCR test at TestCenter Danmark, Statens Serum Institut, Copenhagen, Denmark as usual. Besides the planned oropharyngeal swab performed in the test center, the participants will have additional specimens collected in form of saliva, nasopharyngeal-, nasal-, and oropharyngeal swabs. These will all be used for the detection of nucleic acids from the four most common strains of influenza (B Yamagata, B Victoria, A H1N1 and A H3N2), SARS-CoV-2 and RSV A/B. Further we will measure immune mediating cytokines, chemokines, and interleukins in the different specimens. These analyses will be performed at Technical University of Denmark (DTU).

ELIGIBILITY:
The inclusion criterion:

A. 18 years or more of age requiring a test for COVID-19.

The exclusion criteria are :

A. Neck breathers (tracheostomy/laryngectomy patients) or other nasopharyngeal or oropharyngeal anomalies that do not allow for sampling using swabs.

B. Do not understand oral or written Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
RT-PCR for upper airway viral diagnostics | 1 day
  the detection of nucleic acids from the four most common strains of influenza (B Yamagata, B Victoria, A H1N1 and A H3N2), SARS-CoV-2 and RSV A/B

SECONDARY OUTCOMES:
local immunological mediators from the upper airway tract | 1 day
  measure interferon γ (IFN-γ), C-X-C motif chemokine 10 (CXCL10/IP10), interleukin 10 (IL-10), interleukin 12p70, interleukin 13 (IL-13), interleukin 1β (IL-1β), interleukin 2, interleukin 4 (IL-4), interleukin 5 (IL-5), interleukin 6, CXCL8, tumor necrosis factor α (TNF-α), C-C motif chemokine 5 (CCL5/RANTES), interferon α2a, and granulocyte macrophage colony-stimulating factor (GM-CSF).

CONTACTS AND LOCATIONS:
Locations (1):
- Valby COVID19 testcenter, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Lopez-Perez M, Benfield T, Jakobsen KK, Dal MH, Stange SD, Ersboll AK, Larsen H, Berger SS, Gredal T, Buchwald Cv, Kirkby N, Todsen T. Diagnostic performance of upper airway sampling sites for SARS-CoV-2 and influenza testing. Microbiol Spectr. 2026 Jan 6;14(1):e0221225. doi: 10.1128/spectrum.02212-25. Epub 2025 Nov 17. PMID 41247054